CLINICAL TRIAL: NCT02652884
Title: Evaluation of Potential Benefits of Using Steroids in the Postoperative Transient Hypoparathyroidism Total Thyroidectomy
Brief Title: Steroids in the Postoperative Transient Hypoparathyroidism Total Thyroidectomy
Acronym: Corthyroid
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2627
Record Dates: First submitted 2016-01-05; First posted 2016-01-12 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-01

CONDITIONS: Transient Hypoparathyroidism
Keywords: transient hypoparathyroidism; steroids; total thyroidectomy
MeSH Terms: interventions — Phosphates; betamethasone acetate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): will receive single dose intramuscular corticosteroid deltoid deposit (as phosphate and betamethasone acetate, 2 mL) for immediate postintubation.
  Interventions: Drug: phosphate and betamethasone acetate, 2 mL.
- Group 2 (Placebo Comparator): will receive 2 ml saline 0.9% NaCl in deltoid immediately postintubation.
  Interventions: Drug: saline 0.9% NaCl

INTERVENTIONS:
Drug: phosphate and betamethasone acetate, 2 mL. — single dose of intramuscular depot corticosteroid
  Other Names: cronodose
  Arms: Group 1
Drug: saline 0.9% NaCl — single dose of intramuscular placebo
  Other Names: placebo
  Arms: Group 2

SUMMARY:
The incidence of thyroid cancer (TC) has increased exponentially worldwide. The increase in diagnosed cases brings about an increase in the number of surgeries performed on the thyroid gland, especially total thyroidectomy (TT), given that at present is still the gold standard of treatment.

Transient postoperative hypoparathyroidism (HPT) is one of the most frequent complications, with an incidence of between 10 and 46% according to different sources. HPT involves longer hospital stay, serial measurements of blood glucose, treatment with calcium and vitamin D (with potential risk of hypercalcemia) and therefore an increase in terms of the costs of the health system.

While the investigators know the analgesic, anti-inflammatory, immunomodulatory and anti emetic of corticosteroids in thyroid surgery, the literature available to date is discordant in the use of steroid and its interaction with the HPT making clear the need for randomized clinical trials specific to analyze these variables more accurately.

As inflammation and edema constitute a proposed surgical manipulation in the pathogenesis of HPT component, investigators decided t conduct a prospective randomized, triple-blind, in order to assess the potential benefits of the most common postoperative complication reported in TT.

Our primary objective is to evaluate the safety and efficacy of single-dose corticosteroids deposit immediately postintubation in preventing the development of transient hypoparathyroidism (PTH, serum calcium and symptoms) in patients after TT.

DETAILED DESCRIPTION:
Triple-blind randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

* adult
* thyroidectomy postoperative
* prepaid affiliate patients

Exclusion Criteria:

* allergy
* CKD
* idiophatic thrombocytopenic purpura
* hyperthyroidism
* chronic use of corticoids
* no follicular cancer, nonpapillary
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative Hypocalcemia | 3 days
  Serial postoperative blood samples will be made to detect hypocalcemia (defined as <8,5 mg/dL)
  1. at 1 hour postoperative from skin closure,
  2. at 6 hours after surgery
  3. 24 hours
  4. 72 hours

SECONDARY OUTCOMES:
Related Adverse Events | 30 days
  Any negative effects of corticosteroids will be also recorded in the postoperative and during 30 days follow up after surgery.
  Major side effects associated with glucocorticoid therapy are:
  Gastrointestinal (Gastritis, Peptic ulcer disease, Pancreatitis, Steatohepatitis, Visceral perforation) Dermatologic and soft tissue (Skin thinning and purpura) Cardiovascular (Arrhythmias, Hypertension, Hypotension)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Achaval, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Figari Marcelo, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided